CLINICAL TRIAL: NCT05921344
Title: Preclinical Research of Multi-channel Microspatial Offset Raman Scattering Spectroscopy (mμSORS) for Noninvasive Blood Glucose Detection
Brief Title: Preclinical Research of mμSORS for Noninvasive Blood Glucose Detection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Shanghai Photonic View Technology Co., Ltd. (Unknown)
Responsible Party: Principal Investigator, Wang Weiqing, Professor, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CCEMD2023001
Record Dates: First submitted 2023-06-19; First posted 2023-06-27 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Type 2 Diabetes; Medical Device
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Preclinical Research of mμSORS for Noninvasive Blood Glucose Detection (Experimental): Enrolled subjects will perform oral glucose tolerance test. A measurement session of blood glucose consists of plasma sample and a measurement by mμSORS will be conducted synchronously.
  Interventions: Device: Multi-channel Microspatial Offset Raman Scattering Spectroscopy (mμSORS) for Noninvasive Blood Glucose Detection

INTERVENTIONS:
Device: Multi-channel Microspatial Offset Raman Scattering Spectroscopy (mμSORS) for Noninvasive Blood Glucose Detection — Blood glucose of participants were measured by venous plasma and multi-channel microspatial offset Raman scattering spectroscopy (mμSORS). The two measurements were collected synchronously and analyzed.

SUMMARY:
This is a single-center, open-label, prospective study. Blood glucose was measured at different time points during oral glucose tolerance testing in patients with type 2 diabetes mellitus, using both venous plasma and multi-channel microspatial offset Raman scattering spectroscopy (mμSORS). Venous plasma glucose was set as gold standard.The two measurements were collected synchronously so as to calculate the mean absolute relative difference (MARD) and the consensus error grid (CEG). Accuracy of non-invasive blood glucose testing by mμSORS will be validated. MARD for two measurement methods in different blood glucose ranges and the safety outcomes of mμSORS such as adverse events will also be assessed.

DETAILED DESCRIPTION:
In order to clinically verify the accuracy and safety of non-invasive blood glucose measurement by the mμSORS technology, and to explore the feasibility of non-invasive detection in multi-indicators of mμSORS, this study will conduct an oral glucose tolerance test on patients with type 2 diabetes. There will be 12 collection points of blood samples as follows: 0-min and post glucose-load 15-min，30-min，45-min，60-min，75-min，90-min，105-min，120-min，135-min，150-min， and 180-min. Approximately 4ml of whole blood was collected at each time point for venous plasma glucose and serum insulin measurement. The blood glucose value measured by mμSORS will be obtained synchronously at the above 12 time points.

ELIGIBILITY:
Inclusion Criteria:

* 1. Subjects with type 2 diabetes mellitus;
* 2. Age ≥ 18 years;
* 3. There are no scars, obvious pigmentation and other factors that interfere with the detection of the palm skin to be tested;
* 4. Fully understand the nature, significance, possible benefits, possible inconveniences or potential risks of this research, and should also understand the research procedures, be willing to complete the entire research process, and provide written consent form.

Exclusion Criteria:

* 1. Type 1 diabetes, monogenic diabetes, pancreatic damage, or secondary diabetes of other causes should be excluded;
* 2. Severe structural heart disease, such as congenital heart disease, rheumatic heart disease, hypertrophic or dilated cardiomyopathy, chronic congestive heart failure (NYHA≥III); acute myocardial infarction within 12 months before enrollment; history of severe liver or kidney dysfunction(MDRD eGFR< 60 ml/min/1.73m2); and mental disorders, etc.;
* 3. With a history of acute complications of diabetes within 3 months before enrollment; or severe chronic complications of diabetes;
* 4. Alcohol dependency or drug abuse;
* 5. Those who have participated in clinical trials of other drugs within 3 months before screening (since the last visit of the previous trial);
* 6. Pregnancy or lactation period;
* 7. Difficulty in venous blood collection or blood-injection-injury phobia;
* 8. Other circumstances that the investigator considers inappropriate to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2023-07-11 (Actual); Primary Completion 2023-09-19 (Actual); Study Completion 2023-10-10 (Actual)

PRIMARY OUTCOMES:
Mean absolute relative deviation (MARD) of venous plasma glucose and glucose values measured by mμSORS at each time point of OGTT. | Four months.
  Glucose will be measured using both intravenous sampling (plasma) and multi-channel microspatial offset Raman scattering spectroscopy (mμSORS) detection synchronously.
Consensus Error Grid (CEG) for venous plasma glucose and glucose values measured by mμSORS at each time point of OGTT. | Four months.
  Glucose will be measured using both intravenous sampling (plasma) and multi-channel microspatial offset Raman scattering spectroscopy (mμSORS) detection synchronously.

SECONDARY OUTCOMES:
MARD for two measurement methods in different blood glucose ranges. | Four months.
  Plasma glucose ranges 3.9-10.0 mmol/L, <3.9 mmol/L and >10.0 mmol/L.
Incidence of Treatment-Emergent Adverse Events | Four months.
  Safety outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Weiqing Wang, Dr., Principal Investigator — Ruijin Hospital
Locations (1):
- Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China